CLINICAL TRIAL: NCT00036556
Title: A Phase III, Randomized Study of Atrasentan in Men With Non-Metastatic, Hormone-Refractory Prostate Cancer
Brief Title: Study of Atrasentan in Men With Non-Metastatic, Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M00-244; NCT00026455 (obsolete NCT alias)
Record Dates: First submitted 2002-05-10; First posted 2002-05-13 (Estimated); Last update posted 2007-08-15 (Estimated); Status verified 2007-08

CONDITIONS: Prostatic Neoplasms
Keywords: Hormone-Refractory Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Atrasentan

INTERVENTIONS:
Drug: Atrasentan

SUMMARY:
This study is being done to evaluate the safety and efficacy of atrasentan in men with non-metastatic hormone-refractory prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with prostate cancer.
* Have a rising PSA while on hormone therapy or following surgical castration.

Exclusion Criteria:

* Have evidence of distant metastatic disease on screening bone scan or CT scan.
* Have received cytotoxic chemotherapy.
* Have received opioid or narcotic medications (such as codeine or morphine) or radiation for pain caused by your prostate cancer in the last 6 months.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 941 (Actual)
Dates: Start 2001-06

PRIMARY OUTCOMES:
Time-to-disease progression will be determined by the time to onset of the earliest of one of the following events: New skeletal lesions, new metastatic extra-skeletal lesions, or an event due to metastatic prostate cancer. | Every 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary Gordon, M.D., Study Director — Abbott
Locations (234):
- United States (94):
  - Urology Centers Of Alabama, Homewood, Alabama
  - Alaska Clinical Research Center, LLC, Anchorage, Alaska
  - Advanced Clinical Trials, Tucson, Arizona
  - Arkansas Urologial Associates, PA, Little Rock, Arkansas
  - Robin V. Smith, MD, Chula Vista, California
  - Urology Associate Of Central California, Fresno, California
  - South Valley Medical Plaza, Gilroy, California
  - San Diego Urology Center, La Mesa, California
  - South Orange County Medical Research Center, Laguna Hills, California
  - UCLA School of Medicine, Los Angeles, California
  - VA Palo Alto, Palo Alto, California
  - Hillcrest Urological Medical Group, Inc., San Diego, California
  - Urology Associates Of San Luis Obispo, San Luis Obispo, California
  - Pacific Clinical Research, Santa Monica, California
  - Western Clinical Research, Inc., Torrance, California
  - Urology Associate, Pc, Denver, Colorado
  - South Fl Medical Research, Aventura, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Dattoli Cancer Center, Sarasota, Florida
  - Urology Treatment Center, Sarasota, Florida
  - Southeastern Urological Center, P.A., Tallahassee, Florida
  - Peachtree Hematology/Oncology Consultants, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Sandy Springs Urology, Atlanta, Georgia
  - Atlanta Va Medical Center, Decatur, Georgia
  - Dreyer Medical Clinic, Aurora, Illinois
  - Northwestern University Medical School, Chicago, Illinois
  - Progressive Care, S.C., Chicago, Illinois
  - Christopher Ryan, MD, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Evanston Hospital Kellogg Cancer Center, Evanston, Illinois
  - Welborn Clinic, Evansville, Indiana
  - Welborn Clinic -East, Evansville, Indiana
  - Urologic Associates, Pc, Davenport, Iowa
  - Iowa Urology, Des Moines, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - Regional Urology, Shreveport, Louisiana
  - LSUHSC, Shreveport, Louisiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Drs. Werner, Murdock, & Francis, Pa Urology Assoc., Greenbelt, Maryland
  - Mid Atlantic Clinical Research, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Michigan Medical Urology, Grand Rapids, Michigan
  - Michigan Institute Of Urology, Pc, Saint Clair Shores, Michigan
  - Lakeside Urology, PC, Saint Joseph, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The Medical Oncology Group, Gulfport, Mississippi
  - Mississippi Center For Clinical Research, LLC, Jackson, Mississippi
  - St. Joseph Oncology, Saint Joseph, Missouri
  - Washington University, St Louis, Missouri
  - Billings Oncology Associates, Billings, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Urology Associate, Reno, Nevada
  - UNM Medical Center, Albuquerque, New Mexico
  - Albany Medical Center South Clinical Campus, Albany, New York
  - HemOnCare, PC, Brooklyn, New York
  - Beth Israel Medical Center, New York, New York
  - NYU Medical Center, New York, New York
  - Nyack Hospital, Nyack, New York
  - The University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - Mckay Urology, Charlotte, North Carolina
  - Urology Specialists Of The Carolinas, Charlotte, North Carolina
  - The Urology Center, Greensboro, North Carolina
  - University Of Cincinnati Medical Center, Cincinnati, Ohio
  - Urologic Specialists Of Oklahoma, Inc., Tulsa, Oklahoma
  - Oregon Urology Specialists, Eugene, Oregon
  - Urologic Associates of Allentown, Allentown, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Urological Associates Of Lancaster, Lancaster, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University Of Pittsburgh, Pittsburgh, Pennsylvania
  - Center for Urologic Care, West Reading, Pennsylvania
  - Multimed Research, Providence, Rhode Island
  - University of TN - Memphis, Memphis, Tennessee
  - Urology Associates, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dept of Veteran's Affairs North Texas Healthcare System, Dallas, Texas
  - Ntouch Research Corporation, Dallas, Texas
  - The University Of TX SW Medical Center At Dallas, Dallas, Texas
  - Uthscsa, San Antonio, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Anthony Middleton, M.D., Salt Lake City, Utah
  - Western Urological Clinic, Salt Lake City, Utah
  - University Of Vermont, Burlington, Vermont
  - Virginia Urology Center, Richmond, Virginia
  - Seattle Urological Associates, Seattle, Washington
  - University Of Washington School Of Medicine, Seattle, Washington
  - Jeffrey Frankel, M.D., Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Midwest Research Specialists, LLC, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Wyoming Research Foundation, Cheyenne, Wyoming
- Australia (8):
  - Prince Of Wales Hospital, Randwick, New South Wales
  - Westmead Public Hospital, Westmead, New South Wales
  - Royal Brisbane Hospital, Herston, Queensland
  - Repatriation General Hospital, Daws Park, South Australia
  - Peter Maccallum Cancer Institute, East Melbourne, Victoria
  - Bayside Urology, Mentone, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Princess Alexandra Hospital, Woolloongabba
- Austria (2):
  - A. Ö. Krankenhaus Mistelbach, Mistelbach
  - Klinik fur Urologie der Universitat Wien, Vienna
- Belgium (7):
  - A.Z. Middelheim, Antwerp
  - A Z St Jan, Bruges
  - University Hospital Erasme, Brussels
  - Uz Gent, Ghent
  - Private Practice Dr.Vekemans, Hasselt
  - C.H.U. Liege, Liège
  - St-Elisabeth Ziekenhuis, Turnhout
- Canada (32):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Wilson Urology, Kelowna, British Columbia
  - Dr. Cal Andreou, Surrey, British Columbia
  - Vancouver Hospital & Health Sciences Centre, Vancouver, British Columbia
  - Dr. P. J. Pommerville, Inc., Victoria, British Columbia
  - Dr. Gary Steinhoff, Clinical Research, Victoria, British Columbia
  - Abbott Clinic, Winnipeg, Manitoba
  - Professional Corporation, Fredericton, New Brunswick
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Valley Professional Centre, Kentville, Nova Scotia
  - The Male Health Centres, Barrie, Ontario
  - The Urology Resource Centre, Burlington, Ontario
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - Hamilton & District Urology Association, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Probidity Medical Research, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Quest Clinical Trials, Markham, Ontario
  - Walk-In Clinic, North Bay, Ontario
  - Jack Barkin, M.D., North York, Ontario
  - The Male Health Centres, Oakville, Ontario
  - Ottawa Hospital Civic Campus, Ottawa, Ontario
  - Advanced Male Fertility Clinic, Scarborough Village, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Service Radio-Oncologie, Chus, Fleurimont, Quebec
  - Hopital Notre-Dame, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Ultramed, Pointe-Claire, Quebec
  - Chuq Pavillon Hotel-Dieu, Québec, Quebec
  - Peter Lau, MD, Saskatoon, Saskatchewan
- France (11):
  - Hôpital Cochin, Paris, Cedex 14
  - Hopital Intercommunal, Créteil, Cedex
  - Hôpital Salvator, Marseille, Cedex
  - Hôpital Pasteur, Nice, Cedex
  - Hôpital Saint Louis, Paris, Cedex
  - Centre Hospitalier Rene Dubos, Pontoise, Cedex
  - Hopital De Pontchaillou, Rennes, Cedex
  - Hopital De Rangueil, Toulouse, Cedex
  - Hôpital D´Auxerre, Auxerre
  - Hôpital Henri Mondor, Créteil
  - Hopital Bichat Claude Bernard, Paris
- Germany (12):
  - Allgemeines Krankenhaus Urologie, Celle
  - Universitätsklinikum Urologie, Essen
  - Universitätsklinkum, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Allgemeines Krankenhaus Barmbek, Hamburg
  - Klinik Und Poliklinik für Urologie und Kinder, Homburg / SAAR
  - Universitätsklinikum Lübeck Urologie, Lübeck
  - Universitätsklinikum Mannheim, Mannheim
  - Urologische Klinik Und Poliklinik Grosshadern, München
  - Klinikum Rechts Der Isar, München
  - Universitat Ulm, Ulm
  - Klinikum Wuppertal GmbH, Wuppertal
- Greece (3):
  - 'Alexandra' Hospital, Athens
  - Pe.Pa.G.N.I Hospital, Heraklion
  - G. Genimatas Hospital, Thessaloniki
- Ireland (3):
  - Tallaght Hospital, Dublin
  - St Vincent'S Hospital, Dublin
  - Mater Misericordiae Hospital, Dublin
- Italy (6):
  - Clinica Urologica I - Università di Bari, Bari
  - Istituto Nazionale per la Ricerca sul Cancro -IST, Genoa
  - Istituto Europeo di Oncologia, Milan
  - Clinica Urologica - Università Di Milano, Milan
  - Istituto di Urologia, Padua
  - Policlinico G. B. Rossi, Verona
- Netherlands (6):
  - Amc, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Medisch Spectrun Twente, Enschede
  - Atrium Heerlen, Heerlen
  - University Hospital Rotterdam, Rotterdam
  - St Franciscus Gasthuis, Rotterdam
- New Zealand (2):
  - Canterbury Urology Research Trust, Christchurch
  - Promed Urology Ltd., Tauranga
- Poland (6):
  - Samodzielny Publiczny ZOZ, Bydgoszcz
  - Katedra i Klinika Urologii - Akademia Medyczna w Gdansku, Gdansk
  - Specjalistyczny Szpital Urologiczny, Katowice
  - Szpital Kliniczny Dzieciatka Jezus, Warsaw
  - Instytut im. Marii Sklodowskiej-Curie, Warsaw
  - Akademia Medyczna we Wroclawiu, Wroclaw
- South Africa (7):
  - Mediclinic Hospital, Petermaritzburg, 3201
  - University Of Stellenbosch, Cape Town
  - University Of Natal - Nelson R Mandela School of Medicine, Durban
  - Kenridge St Joseph Wingl, Parktown
  - Medi-Clinic Hospital, Pietermaritzburg
  - Medical Centre, Pietermaritzburg
  - Pretoria Urology Hospital, Pretoria
- Spain (9):
  - Hospital Juan Canalejo, A Coruña
  - Hospital de la Ribera, Alcira (Valencia)
  - Hospital Vall D'Hebron, Barcelona
  - Hospital de Galdakao, Galdakao-Vizcaya
  - Clinica Puerta De Hierro, Madrid
  - Hospital 12 De Octubre, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Marques De Valdecilla, Santander
  - Instituto Valenciano De Oncologia, Valencia
- Sweden (6):
  - Sahlgrenska University Hospital, Gothenburg
  - Linkoping University Hospital, Linköping
  - Lund University Hospital, Lund
  - Malmo University Hospital MAS, Malmo
  - Karolinska Hospital, Stockholm
  - Uppsala University Hospital, Uppsala
- United Kingdom (20):
  - Royal Devon And Exeter Hospital, Exeter, Devon
  - Lister Hospital, Stevenage, Hertfordshire
  - Northwick Park Hospital, Harrow, Middlesex
  - Western General Hospital, Edinburgh, Scotland
  - Taunton And Somerset Hospital, Taunton, Somerset
  - The Institute Of Cancer Research - Royal Marsden Hospital, Sutton, Surrey
  - St Lukes Hospital, Bradford, West Yorkshire
  - Clatterbridge Centre For Oncology, Bebington, WIRRAL
  - Southmead Hospital, Bristol
  - Addenbrookes Hospital, Cambridge
  - St Richard'S Hospital, Chichester
  - Leighton Hospital, Crewe
  - Gartnavel General Hospital, Glasgow
  - Glasgow Royal Infirmary, Glasgow
  - St Batholomew'S Hospital, London
  - Royal Free Hospital, London
  - Clinical Research Centre - St Georges Hospital, London
  - Hope Hospital, Salford
  - Royal Hallamshire Hospital, Sheffield
  - Southampton General, Southampton